CLINICAL TRIAL: NCT07211256
Title: Efficacy of Home-delivered Transcranial Direct Current Stimulation (tDCS) of the Motor Cortex in Patients With Chronic Pain Transiently Relieved by Motor Cortex rTMS : a Pragmatic Randomized Double Blind Sham Controlled Trial
Brief Title: Efficacy of Home-delivered Transcranial Direct Electrical Stimulation or Chronic Pain
Acronym: Homestim-DC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, Coordinator, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-A02797-38
Record Dates: First submitted 2024-11-11; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Pain; Nociplastic Pain
Keywords: randomized; neuropathic pain; nociplastic pain; placebo controlled; tDCS; home-delivered
MeSH Terms: conditions — Neuralgia; Nociplastic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Active Comparator): Active tDCS of the motor cortex
  Interventions: Device: tDCS of the motor cortex
- Sham tDCS (Sham Comparator): Sham tDCS of the motor cortex
  Interventions: Device: tDCS of the motor cortex

INTERVENTIONS:
Device: tDCS of the motor cortex — Home-delivered tDCS device

SUMMARY:
This clinical investigation aims to evaluate the efficacy and safety of a home-based device providing electrical stimulation of the brain named transcranial direct current stimulation (tDCS ) , in patients with chronic pain who have been transiently relieved by repetitive transcranial magnetic stimulation delivered at hospital (less than one month benefit). The general objective is to show that these patients may best benefit from home based tDCS while rTMS performed in hospital has only limited and transient efficacy. Each participant will be randomized into one of two arms to receive during 3 months either active tDCS or sham tDCS. Neither the investigator nor the patient will be aware of the treatment. The efficacy will be assessed on pain intensity (primary outcome at 3 months) and several secondary outcomes (qualify of life, pain symptoms , global impression of change, pain relief, sleep, anxiety, depression) every month for up to 3 months. Safety will be assessed at each follow up visit for up to 3 months. The participants will be asked to self stimulate themselves with the device 5 days per week for about 20 minutes.

DETAILED DESCRIPTION:
This will be a randomised, double-blind, parallel-group, bi-centric study versus placebo stimulation. Patients undergoing previous treatment with rTMS of the motor cortex in routine in our pain center and with at least 30 % pain relief with rTMS (after 10 sessions) but only transient pain relief (less than one month) will stop their treatment for at least one month. They will then be randomised to receive one of the 2 treatments under study (active tDCS of the motor cortex, placebo tDCS of the motor cortex, TENS eco plus). The protocol will involve a 20-minute tDCS session (2 mA) at home, 5 days a week for 12 weeks. The treatment will continue for 12 weeks and the final evaluation will take place at 12 weeks.

TENS ECO PLUS is a portable transcranial direct current stimulation (tDCS) system (tDCS kit) supplied by the Monath Electronic laboratory, designed for use at home; this system will first be tested in hospital during a test session with explanations to the patient on how to use it. The stimulation intensity is blocked above a certain threshold by the system to avoid any risk of epileptic seizure. Sham or placebo stimulation uses the same medical device without active stimulation.

Given the exploratory nature of the trial and in order to reduce study participant's exposure to a potentially useless treatment, blinded interim analysis will be conducted dring the course of the trial in the first 40 enrolled patients and the study will be stopped early if this analysis suggests large differences between the two treatment groups or conversely shows obvious futility.

ELIGIBILITY:
Inclusion Criteria:

Chronic pain for at least 6 months Pain intensity ≥ 4/10 on 0-10 NRS Pain present every day or nearly every day Neuropathic pain (DN4 score ≥ 4/10) or nociplastic pain (Kosek et al Pain 2021) Patients previously treated with rTMS of the motor cortex in routine in our pain center but with only transient efficacy (ie, efficacy for less than one month, defined as pain intensity improved by at least 30 %) Affilitated to social security

Exclusion Criteria:

Contraindications to tDCS as stated in the manufacturer brochure (ie, implantable device , severe cognitive disorders, epilepsia, skin problems where will placed the electrodes, arterial or venous thrombosis, thrombophlebitis, metallic intracranial implant, cranioth-omy, incracranial aneuvrysm, cerebral tumor, severel sleep disorders such as narcolepsia) Conciomitant treatment which might increase the risk of epilepsia such as high doses opioids (≥ 140 mg morphine equivalent) or high. doses tricyclic antidepressants (≥ 150 mg per day) Pregnancy or lactation Age below 18 or > 80 years Pending litigation related to pain Pain more severe than neuropathic or nociplastic pain requiring treatment Severe disease such as cancer Severe psychiatric condition (psychosis) Impossible to be followed for up to 3 months Participation in a recent protocol (less than 3 months) Psychoactive drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Self reported pain intensity in a diary | Baseline and 12 weeks
  Weekly average of the last 7 numerical pain scores (from 0 no pain to 10 maximal pain imaginable) recorded every day by the patient at the end of the treatment as compared to baseline values

SECONDARY OUTCOMES:
Effects on self reported pain intensity over the course of the study | over the course of the study from baseline to week 12
  Weekly averaged pain intensity on numerical pain scales (0-10, with 0 no pain and 10 maximal pain imaginable) self reported on pain diary over the course of the study
EQ-5D-5L (EuroQol) | Baseline, then week 1 (± 3 days), week 4, week 8 and week 12
  Quality of life on EQ-5D-5L scale including 5 levels of perceived problems each rated on 0-3 categorical scales
Brief Pain Inventory | Baseline, then week 1 (± 3 days), week 4, week 8 and week 12
  Average pain on numerical pain scales (from O no pain to 10 maximal pain) on the Brief Pain Inventory (BPI)
Neuropathic Pain Symptom Inventory (NPSI) | Baseline, then week 1, week 4, week 8 and week 12 after the treatment
  Self reported neuropathic pain questionnaire to assess 5 neuropathic dimensions rated on the same numerical rating scales (from 0 no symptom to 10 maximal symptom). This questionnaire will be proposed only for neuropathic patients.
Fibromyalgia Impact Questionnaire (FIQ) | Baseline, then week 1 (± 3 days), week 4, week 8 and week 12
  Self reported questionnaire assessing the impact of fibromyalgia on everyday life. This questionnaire will only be proposed to patients with fibromyalgia.
Hospital anxiety and depression scale (HADS) | Baseline, then week 1 (± 3 days), week 4, week 8 and week 12
  Symptoms of anxiety rated on 21 on the HADS with 0 indicating no anxiety and 21 indicating the maximal level of anxiety
Medical outcomes study sleep scale (MOS sleep) | Baseline, then week 1 (± 3 days), week 4, week 8 and week 12
  Sleep impairement on the MOS sleep allowing to calculate two indexes (sleep problem index 6 and 9)
McGill pain questionnaire short form (SF-MPQ) | Baseline, then week 1 (± 3 days), week 4, week 8 and week 12
  SF-MPQ (Melzack et al 1986) allowing to evaluate the sensory and affective dimension of pain; the sensory dimension of pain is rated on 30 with 30 indicating more severe sensory dimension of pain
Pain Catastrophizing Scale (PCS) | Baseline then 1 week ± 3 days then 4 weeks, 8 weeks and 12 weeks
  Pain catastrophizing on the PCS (Sullivan et al), scored from 0 to 52 (with 52 indicating worse catastrophizing)
Patient global impression of change (PGIC) | Baseline then 4 weeks, 8 weeks and 12 weeks
  PGIC as assessed on a 7 category scale from much improved to much deteriorated
Treatment-emergent adverse effects of home delivered tDCS | Every day over the course of the study and at each follow up visit, at days 3 (initial follow up safety visit) then days 10, week 4, week 8 and week 12
  Treatment emergent adverse effects will be assessed at each follow up visit by the investigators. Patients will also report any adverse effect occurring immediately after each session of tDCS or between sessions on a self diary.
Categorical pain scale | Baseline then 10 days (± 3 days), 4, 8 and 12 weeks
  Categorical pain scale (from no pain to very severe pain)
Blinding assessment | 12 weeks
  A blinding assessment as used in our prior studies will be proposed to every patient including 2 questions : what treatment they think they had received (active or placebo) ; the main reason for their choice (efficacy, side effects, both, other reasons)
Satisfaction with the treatment | 12 weeks
  Satisfaction with the treatment will be assessed on a 0 to 10 numerical scale (0 = not satisfied ; 10 : extremely satisfied)
Interference score of the Brief Pain Inventory | Baseline then 1 week, 4 weeks, 8 weeks and 12 weeks after the treatment
  Interference score rated from 0 to 70 from the Brief Pain Inventory
Pain as its least from the Brief Pain Inventory | Baseline then 1 week, 4 weeks, 8 weeks and 12 weeks after the treatment
  Pain intensity as its least over the past 24 hours rated on a numerical rating scale from 0 to 10
Pain as its worst from the Brief Pain Inventory | Baseline then 1 week, 4 weeks, 8 weeks and 12 weeks
  Pain intensity as its worst over the past 24 hours rated on a 0-10 numerical rating scale
Clinician global impression of change (CGIC) | Baseline and at 12 weeks
  7 category Clinician based global impression of change from severe deterioration to significant improvement
EQ5D -5L Euroqol Visual analog scale | Baseline, week. 1, weeks 4, weeks 8 and weeks 12 after the treatment
  Visual analog scale rated from 0 to 100 to measure health status with 0 being the worse health status and 100 being the best possible health status
Symptoms of depression on the Hospital Anxiety and Depression Scale (HADS) | Baseline then one week, 4 weeks, 8 weeks and 12 weeks
  Symptoms of depression rated on 21 on the HADS with 0 indicating no anxiety and 21 indicating the maximal level of depression
Short Form McGill Pain Questionnaire SF-MPQ | Baselinen one week, 4 weeks, 8 weeks and 12 weeks after the treatment
  SF-MPQ allowing to evaluate the affective dimension of pain; the affective dimension of pain is rated from 0 to 12 with 12 indicating more severe sensory dimension of pain

OTHER OUTCOMES:
Predictors of the response to tDCS | Baseline
  Clinical predictors of the response to tDCS will be assessed based on multivariate analyses taking into account the patients profiles at baseline
Easyness of use | Days 3-5, then week 1, then weeks 4, 8 and 12 after the treatment
  Patients will be questioned at each time point over the course of the study about the easyness of use of the home based device, whether they experienced difficulty and which were they. These will be assessed by open questions only.
Predictor of the response to placebo | Baseline
  A specific questionnaire will be used to assess the risk of placebo response

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, MD PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Centre d'Evaluation et de Traitement de la douleur, INSERM U 987, Boulogne-Billancourt, Hauts de Seine, France

IPD SHARING:
Plan to Share IPD: No
Problem of confidentiality